CLINICAL TRIAL: NCT01962142
Title: Subjective and Objective Assessment of Activity Limitation in Asthma Patients
Brief Title: Assessment of Activity Limitation in Asthma Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Other Study IDs: B076201214059
Record Dates: First submitted 2012-10-15; First posted 2013-10-14 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2015-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Exacerbated asthma patients
  Interventions: Other: Assessment of activity capacities

INTERVENTIONS:
Other: Assessment of activity capacities

SUMMARY:
Limitation of activity is one of the main item used by composites scores designed to assess the level of asthma control. Since this item is systematically subjectively assessed by the patient, the investigators would like to know if these subjective data are correlated with objective data.

Aims of this study are: 1) To describe what means "limitation of activity" for asthma patients and how they deal with; 2) To describe the objective exercise capacity and characteristics of daily activity in two situations (on exacerbation, out of an exacerbation).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma made by a pulmonologist.
* Age ≥ 18 yrs-old, < 65 yrs-old.
* Moderate or severe exacerbation of asthma (as defined by Reddel et al in 2009) at the time of inclusion.

Exclusion Criteria:

* All other diseases than asthma that can affect the physical activity (e.g. orthopaedic or neuromuscular disease, cardiac or vascular disease).
* Pregnancy or suspicion of pregnancy at the time of inclusion. The women who become pregnant during the study period will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Exacerbated asthma patients coming to the outpatient clinic of pulmonology.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Energy expenditure (expressed in MET's) measured during an ergospirometry, at the time of an exacerbation of asthma and 6 weeks later. | At the time of inclusion
  One MET (Metabolic Equivalent of Task) is equal to an oxygen uptake about 3.5 ml O2/kg/min.

SECONDARY OUTCOMES:
Walking distance in 6 min (expressed in meters) measured at the time of an exacerbation of asthma and 6 weeks later. | 6 weeks
Quality of life (assessed with the Asthma Quality of Life Questionnaire) measured at the time of an exacerbation of asthma and 6 weeks later. | At the time of inclusion
Self-assessment of activity limitation | 7 last days before inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU St Pierre; pulmonology department, Brussels, Belgium